CLINICAL TRIAL: NCT00586092
Title: A Phase I Study of ABT-510 in Combination With Bevacizumab in Advanced Solid
Brief Title: A Phase I Study of ABT-510 in Combination With Bevacizumab in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herbert Hurwitz (Other)
Collaborators: Genentech, Inc. (Industry); Abbott (Industry)
Responsible Party: Sponsor-Investigator, Herbert Hurwitz, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Pro00008797; NCT00276562 (obsolete NCT alias)
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Solid Tumors
Keywords: Phase I; Phase 1; avastin; bevacizumab; ABT-510; solid tumors; angiogenesis
MeSH Terms: interventions — Bevacizumab; NAc-Sar-Gly-Val-(d-allo-Ile)-Thr-Nva-Ile-Arg-ProNEt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): This trial employs a phase I design with a dose escalation stage (stage I) and an expansion stage (stage 2) to better describe the tolerability of this combination and the effect of this combination on several biomarkers. In this second stage there will be two groups, each with ten patients, to better describe the tolerability of the bevacizumab/ABT-510 combination and the effect of this combination on several biomarkers. The primary objective of this study is to estimate the MTD/recommended phase II dose regimen. All other objectives are exploratory in nature.
  Interventions: Drug: bevacizumab, ABT-510

INTERVENTIONS:
Drug: bevacizumab, ABT-510 — * Stage 1 (Cohorts -1, 2, 2, 3) ABT-510: 25, 50, 50, 100 mg SC BID*, bevacizumab: 5, 5, 10, 10 mg/kg IV every 14 days*
  * Stage 2 (RPTD) ABT-510: X mg SC BID**, bevacizumab: Y mg/kg IV every 14 days**
    * Stage I is the dose escalation stage. Stage II will include an additional 20 patients (10 patients in each group) enrolled at the RPTD in two different schedules to better assess safety and biomarker correlates.
      * *Both agents begin on Day 1 of Cycle 1.
        * **At the RPTD, ½ the patients will begin ABT-510 (Dose X) on Day 1 and bevacizumab (Dose Y) on Day 15 and the other ½ of the patients will begin bevacizumab on Day 1 and ABT-510 on Day 15. This will allow for a collection of some preliminary data of wound angiogenesis effects of ABT-510 alone versus the combination and bevacizumab alone versus the combination.
  Other Names: avastin

SUMMARY:
The primary objective of this study is to determine the recommended Phase II dose for the combination of ABT-510 plus bevacizumab in patients with advanced solid tumors and to evaluate dose limiting toxicities and non-dose limiting toxicities of this combination. The secondary objectives are to collect preliminary data on the effect of the combination of ABT-510 plus bevacizumab versus each agent individually on dermal wound angiogenesis in a skin biopsy and to collect preliminary data on the clinical activity of this combination (tumor response rate, progression-free survival, rate of stable disease > 6 months).

DETAILED DESCRIPTION:
ABT-510: In the early 1990s, thrombospondin (TSP-1) was first recognized as an endogenously produced inhibitor of angiogenesis. Since then, thrombospondin has been shown to inhibit neovascularization and tumorigenesis in numerous mouse models. Its anti- angiogenesis properties have been localized to its N-terminal region. Although smaller fragments of this region retain some of thrombospondin's anti-angiogenesis properties, researchers have discovered that specific amino acid substitutions can greatly enhance these properties. From these efforts, ABT-510, a nine-amino acid synthetic peptide has emerged as a novel anti-angiogenesis agent. The peptide is soluble and stable in water and is administered parenterally as an acetate salt in 5% dextrose solution for clinical use.

ABT-510 has been evaluated in three Phase I studies: one single-dose study in healthy volunteers and two studies in cancer patients. Doses ranging from 10 mg to 260 mg have been evaluated as IV infusions (30-minute), subcutaneous bolus injections, or 24-hour subcutaneous infusions. Overall, ABT-510 has been well tolerated. A preliminary review of the 103 case report forms collected to date identified a total of 1306 adverse events. Ninety-one percent (1195/1306) of these events were considered to be mild or moderate in nature. Eighty-one percent (1052/1306) of these events were reported as not related to or probably not related to ABT-510. The most common adverse events, occurring in >10% of the patients, include injection site reaction, asthenia, abdominal pain, nausea, anorexia, pain, headache, vomiting, diarrhea, dyspnea, constipation, cough increased, back pain, peripheral edema, dizziness, insomnia, anemia, fever, sweating, chest pain, and rash.

Bevacizumab (Avastin) is a recombinant, humanized, monoclonal antibody directed against vascular endothelial growth factor (VEGF). This antibody blocks binding of the ligand VEGF with its receptor. VEGF is known to play a pivotal role in tumor angiogenesis and is a significant mitogenic stimulus for arterial, venous, and lymphatic endothelial cells. It can induce vascular permeability essential for extracellular remodeling and can serve as an endothelial cell survival factor. Phase III studies in 1st line colorectal cancer, 2nd line colorectal cancer, 1st line breast cancer, and 1st line non-small cell lung cancer have all demonstrated clinical benefit in terms of overall survival, progression free survival, and tumor response [Refs.. HH NEJM, A Sandler ASCO2005, L Miller ASCO 2005]. Efficacy has also been noted in phase II studies of renal cell, ovarian, glioma, and other tumor types. Side effects of bevacizumab include approximately 10-20% rate of hypertension requiring anti-hypertensives, uncommon aterial thromboembolilc events (myocardial infarction, unstable angina, cerebrovascular events, transient ischemic attacks, etc) with background rates increased from approximately 1-2% to 2-4%, and an approximately 1-2% risk of GI perforation.

Aside from this pivotal phase III colorectal cancer study, the dose of bevacizumab used for all other clinical trials has been 10mg/kg biweekly. A dose of bevacizumab at 10 mg/kg will be used in this study because it is consistent with the dosing used in most ongoing and planned bevacizumab studies and it has been shown, when compared to lower doses, to have comparable or improved activity.

Based on available data, it is a reasonable hypothesis that the combination of ABT-510 and bevacizumab will be a safe and potentially efficacious anti-angiogenesis strategy for the treatment of adult solid tumors. This combination may have utility directly or may prove useful when subsequently combined with other anti-angiogenic agents or standard chemotherapy regimens. An important aspect of this proposed study will be the inclusion of a clinical dermal wound angiogenesis assay which will help quantify and characterize the anti-angiogenic contribution of each agent in this combination. Therefore, this study is meant to provide important safety information on this combination, but also insight into the additive mechanistic effects of two agents with different mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced solid tumor refractory to standard therapy or for whom there is no standard therapy.
* Patients must not have had radiation therapy, hormonal therapy, biologic therapy or chemotherapy for cancer within the 21 days prior to study Day 1. Patients must not have had major surgery within the 28 days prior to study Day 1 or minor surgical procedures within the 14 days prior to study Day 1.
* Age > 18 years.
* ECOG performance status of 0-1 (see Appendix A).
* Patients must have normal organ and marrow function as defined below:

  * hemoglobin > 9.0g/dL; absolute neutrophil count > 1,500/μl; platelets > 100,000/μl; total bilirubin < 1.5 X upper limit of normal (ULN), AST(SGOT)/ALT(SGPT) < 2.5 X ULN, < 5 X ULN if known hepatic metastases; Urine protein:creatinine ratio < 1.0; creatinine clearance > 50 mL/min/1.73 m2; PT/INR/PTT < 1.2X ULN
* The effect of the investigational drugs on the developing human fetus is not known, but these drugs are likely to be embryo- and feto- toxic. Women of child-bearing potential must agree to use adequate contraception (either surgical sterilization; approved hormonal contraceptives such as birth control pills, Depo-Provera, or Lupron Depot; barrier methods such as condom or diaphragm along with spermicide; or an IUD). Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician and study PI immediately. Patients should be willing to use adequate contraception for three months following discontinuation of study drug.
* The patient is able to self-administer or has a caregiver who can reliably administer subcutaneous injections.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had radiation therapy, hormonal therapy, biologic therapy, or chemotherapy for cancer within the 21 days prior to Day 1 of the study. Patients with prostate cancer who are already receiving androgen deprivation therapy (ie. leuprolide or goserelin) for longer than 3 months may continue on this therapy during the study.
* Patients who have received any other investigational agents within the 28 days prior to Day 1 of the study.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis, the uncertain risk of this regimen on tumor bleeding, and because these patients often develop progressive neurological dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with primary malignancies known to metastasize to the brain (such as lung cancer, breast cancer, renal cell cancer, , sarcoma, carcinoma of unknown primary, melanoma, and head and neck cancers) or patients with symptoms of brain metastases should have a brain MRI within 28 days of enrollment to confirm the absence of CNS metastases. Contrast CT is acceptable for patients who are unable to undergo a brain MRI.
* Patients with poorly controlled or clinically significant atherosclerotic vascular disease including CHF NY Heart Class > 2 (see Appendix B); angina requiring nitrates; MI, CVA, TIA, angioplasty, cardiac or vascular stenting in the past 6 months; or ventricular arrhythmia requiring medication.
* History of intolerance of prior treatment with bevacizumab or ABT-510. Prior treatment with these agents is otherwise permitted.
* Poorly controlled hypertension (> 160/100). Initiation or adjustment of BP medication is permitted prior to study entry provided that patient has 3 consecutive BP readings less than 150/90 mmHg each separated by a minimum of 24 hours. These readings should be collected prior to first skin biopsy.
* History of thrombosis within 3 months prior to enrollment or current use of therapeutic anticoagulation. Prophylactic low-dose anticoagulation for indwelling catheters is permitted; PT/PTT must be within normal limits.
* Use of antiplatelet agents other than aspirin (< 325 mg/day) or standard dose NSAIDs.
* Presence of bleeding diathesis, coagulopathy, or major bleeding event such as an acute GI bleed requiring transfusion or invasive intervention or hemoptysis greater than 1 tablespoon within 6 months prior to Day 1 of the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit safety or compliance with study requirements. In addition, patients with non-healing wounds will not be eligible for this study.
* Pregnant women are excluded from this study because the investigational drugs have potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these drugs, breastfeeding should be discontinued if the mother is treated on this study.
* Patients with squamous cell carcinoma of the lung.
* History of intra-abdominal fistula, gastrointestinal perforation or intr-abdominal abscess within 6 months prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To determine the recommended Phase II dose for the combination of ABT-510 plus bevacizumab | Each Cycle (28-days)

SECONDARY OUTCOMES:
To collect preliminary data on the clinical activity of this combination (tumor response rate, progression-free survival, rate of stable disease > 6 months). | Each Cycle (28-days)

CONTACTS AND LOCATIONS:
Overall Officials: Herb Hurwitz, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States